CLINICAL TRIAL: NCT06310811
Title: A Safety, Efficacy, and Pharmacokinetics Study of Anti-CD19 CAR-T Cell Therapy in Participants With Moderate to Severe Active Systemic Lupus Erythematosus
Brief Title: Anti-CD19 CAR-T Cell Therapy in Participants With Moderate to Severe Active Systemic Lupus Erythematosus
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: R&D strategy adjustment
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, MEI HENG, Chief physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD06-04-01
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Safety; Effective
Keywords: CD19 CART, SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: All patients will be treated with RD06-04 cell injections in a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cell injection (Experimental)
  Interventions: Drug: RD06-04 Cells injection

INTERVENTIONS:
Drug: RD06-04 Cells injection — Patient will be treated with RD06-04 cells when enrolled in the study

SUMMARY:
This is an open, Phase I, investigator-initiated study (IIT) to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of RD06-04 in patients with moderate or severe active SLE.

This study will explore the safety of escalating doses of RD06-04 by presetting two dose levels (DL), with 3 to 6 patients enrolled in each dose level. After safety conclusions are reached in each group, the investigator can select the corresponding dose group to expand cases based on treatment response, but the total number of cases will not exceed 12.

This study will enroll patients in a 3+3 design with two DLS: 1×105 CAR+T cells /kg for DL1 and 5×105 CAR+T cells /kg for DL2.

Dose increment Refer to the 3+3 dose increment principle. Three subjects are expected to be enrolled in each dose group.

1. Dose increment should start from the minimum dose, and it is not possible to conduct an incremental study of 2 or more dose groups at the same time.
2. If 1 case of DLT occurs in each dose group, the dose level will be extended to 6 subjects. If 6 subjects at this dose level ≥2 subjects develop DLT, the dose level exceeds the MTD. The previous lower dose level will be extended to 6 subjects, and if 6 subjects have already been enrolled in the previous lower dose level, and only ≤1 of these 6 subjects develop DLT, this lower dose level will be considered MTD.
3. If DLT occurred in ≥2 subjects in the highest dose group, the researcher could select a dose between the high dose group and the medium dose group according to the specific situation and perform MTD evaluation.
4. If the dose increase to the highest dose group still does not reach DLT, researchers can explore the safety and efficacy of higher doses according to specific circumstances.

Case expansion:

After the completion of DLT evaluation in all dose groups, the investigators could select the corresponding dose group of extended cases according to the treatment response, but the total number of cases should not exceed 12 (extended cases were not evaluated by DLT).

ELIGIBILITY:
Inclusion Criteria:

* 1.The subjects voluntarily participated in the experiment and signed the informed consent.

  2. Age ≥18 years old and ≤70 years old, regardless of gender. 3. Diagnosis of SLE according to the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria 2019 or the 2012 International Clinical Collaboration Group on Systemic Erythraeus (SLICC) criteria.

  4. Prior to screening, patients must have been treated with glucocorticoids combined with immunosuppressants and/or biologics for at least 2 months, and the dose is stable for >2 weeks, and the disease is still active (i.e., previous treatment with glucocorticoids + immunosuppressants or glucocorticoids + immunosuppressants + biologics, and any of the above drugs are not eligible for single drug use). Oral corticosteroids must meet the following requirements: 1) Prednisone (or equivalent) ≥7.5mg/ day; 2) There is no minimum daily dose requirement for corticosteroids when used in combination with immunosuppressants and/or biologics.

  5. Screening is positive for antinuclear antibody (ANA), and/or anti-DS-DNA antibody, and/or anti-Smith antibody.

  6. The SLEDAI-2K score in the screening period was >6, and the "clinical" SLEDAI-2K score was ≥4.

Note: "Clinical" SLEDAI-2K is a score in the SLEDAI-2K score that does not include results attributable to any urine or laboratory tests (including immunological indicators) :

7. The BILAG2004 score meets at least one of the following conditions:

a) ≥1 organ system BILAG2004 Class A disease b) ≥2 organ systems BILAG2004 Class B disease 8. Physician General assessment (PGA) score ≥1.0 (0-3 on visual analogue scale VAS) during screening.

9. Organ function and laboratory tests:

1. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST≤3× upper normal limit (ULN), total bilirubin (TBIL) ≤2×ULN (except Gilbert syndrome).
2. Renal function: creatinine ≤1.5×ULN or creatinine clearance ≥40 ml/min.
3. Blood routine: neutrophil count ≥1×109/L, hemoglobin ≥60g/L, platelet count ≥20×109/L, lymphocyte count >0.3×109/L.
4. Coagulation function: International standardized ratio (INR) ≤ 1.5×ULN, or prothrombin time (PT) ≤ 1.5×ULN.
5. Blood oxygen saturation (SpO2) at rest in indoor air ≥92%.
6. Echocardiography showed left ventricular ejection fraction (LVEF) ≥50%. 10. The serum or urine pregnancy test results of fertile female subjects at the time of screening were negative.

   11. Fertile women must consent to the use of highly effective contraceptive methods for contraception from at least 28 days before the start of the infusion until 12 months after the RD06-04 reinfusion. Fertile men must consent to the use of an effective barrier method of contraception from the start of DTP until 12 months after RD06-04 reinfusion, and should not donate semen or sperm throughout the trial period.

   Exclusion Criteria:
   * 1. Combined with other autoimmune diseases, systemic treatment is required. 2. The presence of uncontrolled lupus crises within 8 weeks prior to screening, including acute lupus nephritis, severe neuropsychiatric lupus, severe hemolytic anemia, severe immune thrombocytopenia, agranulophilia, severe heart damage, severe lupus pneumonia, severe lupus hepatitis, and severe vasculitis, was assessed by the investigators as not suitable for participation in this study.

     3. Clinically significant central nervous system diseases or pathological changes not caused by lupus prior to screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, convulsions/convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, cerebral organ syndrome, or psychosis.

     4. Have a history of allogeneic bone marrow or stem cell transplantation or solid organ transplantation (such as kidney, lung, heart, liver) or plan to undergo such transplantation in the future.

     5. Clinically significant cardiovascular dysfunction in the 12 months prior to screening, including but not limited to: Class III or IV heart failure as defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, or any ventricular arrhythmias.

     6. A history of malignant neoplasm within 5 years prior to signing the ICF, with the exception of sufficiently treated or surgically resected non-melanoma skin cancer or carcinoma in situ (e.g. cervical, bladder, breast) with no residual disease.

     7. Pregnant or lactating women. 8. A history of recurrent infections requiring hospitalization and intravenous antibiotics (e.g., 3 or more infections of the same type in the past year).

     9. There are active infections, such as infectious pneumonia and tuberculosis, that need systematic treatment within 2 weeks before the treatment.

     10. Hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA test positive; Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; Human immunodeficiency virus (HIV) antibody positive.

     11. Have received live attenuated vaccine within 4 weeks prior to treatment or plan to receive live attenuated vaccine during the course of the study.

     12. Receiving high doses of corticosteroids (prednisone ≥60 mg/ day or equivalent) within 4 weeks prior to drenching, or failing to taper prednisone to ≤10 mg/ day 5 days prior to drenching.

     13. As indicated in Table 3, tapering or elution of background therapy is not possible prior to eluvial chemotherapy.

     14. Were receiving renal replacement therapy in the 3 months prior to screening or expected to require renal replacement therapy during the study period.

     15. History of drug or alcohol abuse within 1 year prior to screening. 16. History or evidence of suicidal thoughts in the 6 months prior to screening, or any suicidal behavior in the 12 months prior to screening, is considered by the investigator to be a significant risk of suicide.

     17. Use of other study drugs within 4 weeks or 5 half-lives (whichever is older) prior to screening.

     18. A history of hypersensitivity or life-threatening reactions to any ingredient or preparation of an investigational drug or investigational treatment, including chemotherapy. For more information about the ingredients of the investigational drug, see the Investigator's Manual (IB).

     19. Any situation that the investigator believes may affect study participation, pose a safety risk to patients, or may confuse the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-12-03 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | 28 days from cell infusion
The incidence of treatment-based adverse events (TEAEs) and the incidence of serious adverse events (SAEs). | 3 months from cell infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided